CLINICAL TRIAL: NCT01328418
Title: Simultaneous Lengthening of Bilateral Femora and Tibiae in Achondroplastic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilen, Fikri Erkal, M.D. (Individual)
Responsible Party: Mehmet Kocaoglu, MD, Professor, Istanbul Medical School
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Akondroplazi - Bilen
Record Dates: First submitted 2011-04-01; First posted 2011-04-04 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2011-04

CONDITIONS: SHOX Gene With Short Stature
Keywords: Lengthening
MeSH Terms: conditions — Dwarfism

ARMS (1):
- Achondroplasia lengthening (Other)
  Interventions: Procedure: Lengthening over nail

INTERVENTIONS:
Procedure: Lengthening over nail — External fixator is used to lengthen either the femur or the tibia over an intramedullary nail

SUMMARY:
The purpose of this study is to determine whether lengthening of both the tibiae and femora in achondroplastic patients is safe and provides reproducible outcome.

ELIGIBILITY:
Inclusion Criteria:

* Achondroplasia, first lengthening period

Exclusion Criteria:

* Previous lengthening

Ages: 3 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2002-04; Primary Completion 2008-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Paley's functional scoring system | Minimum 2 year follow-up
  Paley's functional scoring system evaluates the results after lengthening or deformity correction procedures: residual limb length discrepancy, any brace or other aid usage, joint contracture, pain, soft tissue dystrophism

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medical School, Istanbul, Turkey (Türkiye)